CLINICAL TRIAL: NCT01985035
Title: Influence of Obstructive Sleep Apnea on Metabolism and Weight Loss in Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Camila Maria de Melo, Msc, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RMR-PRO
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Obstructive Sleep Apnea; Obesity
Keywords: Obstructive sleep apnea; obesity; diet; energy expenditure
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Diet

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Obese Apneic carbohydrate diet (Experimental): Obese apneic individuals will be subject to a energy restriction diet rich in carbohydrates
  Interventions: Behavioral: Diet
- Obese Apneic protein diet (Experimental): Obese apneic individuals will be subject to a energy restricted diet rich in protein
  Interventions: Behavioral: Diet
- Obese Non Apneic carbohydrate diet (Experimental): Obese individuals without Obstructive sleep apnea will be subjected to a energy restricted diet rich in carbohydrates
  Interventions: Behavioral: Diet
- Obese Non Apneic protein diet (Experimental): Obese individuals without Obstructive Sleep Apnea will be subjected to a energy restricted diet rich in protein
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — Reduction of energy intake in order to weight loss
  Other Names: Energy restriction

SUMMARY:
Obstructive sleep apnea (OSA) can impars body weight reduction by changes in body composition and energy expenditure. The objective of this study is to evaluate the influence of OSA in energy metabolism and body mass loss in obese subjects. Ninety obese volunteers of both genders, 45 diagnosed with OSA and 45 without OSA, will be submitted to a dietary intervention of one months. Volunteers will be distributed into four groups: obese OSA PTN with moderate protein diet (1.6 g / kg protein / day), obese OSA CHO diet (0.8 g / kg protein / day) with standard composition diet, obese NSAOS PTN diet moderate in protein and CHO NSAOS obese standard diet. All groups will be instructed to perform a restricted energy diet (less 30% of daily energy expenditure). At baseline and one month after the beginning of the program the following evaluations will be conducted: total energy expenditure measured by doubly labeled water method, resting energy expenditure and thermic effect of food by calorimetry, polysomnography analysis, body composition by pletysmography, food consumption by three days of food diary, blood collection for analysis of lipid profile, visceral proteins, hormones related to control of body weight and inflammation. As hypothesis we believe that apneic obese individuals have greater difficult in weight loss and loss more free fat mass than the obese no apneic and that diets with more protein can contribute to greater weight loss, better body composition and energy expenditure in these population.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 30 and 40 kg/m2;
* Obstructive sleep apnea mild or severe;
* Sedentary.

Exclusion Criteria:

* Intake of any drug that interfere on metabolism such for thyroid or to lose weight;
* Be engaged in other treatment for sleep apnea or obesity;
* Present another sleep disorder;
* Being shift work;
* Present any kind of kidney disease.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-10; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Energy expenditure | up to 4 months
  Measurements of energy expenditure by doubly labeled water for day energy expenditure and by calorimetry for resting energy expenditure and thermic effect of food

SECONDARY OUTCOMES:
Body Composition | Baseline, 1 month, 2 months and 4 months
  Bodu composition evaluation by pletismografy to determine fat mass and fat free mass

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Departamento de Psicobiologia - Universidade Federal de São Paulo, São Paulo, São Paulo
  - Universidade Federal de São Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] de Melo CM, Dos Santos Quaresma MVL, Del Re MP, Ribeiro SML, Moreira Antunes HK, Togeiro SM, Tufik S, de Mello MT. One-month of a low-energy diet, with no additional effect of high-protein, reduces Obstructive Sleep Apnea severity and improve metabolic parameters in obese males. Clin Nutr ESPEN. 2021 Apr;42:82-89. doi: 10.1016/j.clnesp.2020.12.028. Epub 2021 Feb 11. PMID 33745625